CLINICAL TRIAL: NCT04280432
Title: Monocentric Observational Study: Postoperative Pain After Cesarean Section: Incidence and Risk Factors.
Status: Completed | Type: Observational
Sponsor: Instituto de Investigación Hospital Universitario La Paz (Other)
Responsible Party: Sponsor
Other Study IDs: PI-2564
Record Dates: First submitted 2019-09-12; First posted 2020-02-21 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2019-09

CONDITIONS: Chronic Postoperative Pain; Cesarean Section Complications
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cesarean: Women hospitalized for cesarean section
  Interventions: Procedure: CESAREAN

INTERVENTIONS:
Procedure: CESAREAN — Women hospitalized for cesarean section

SUMMARY:
The purpose of this prospective study was to assess chronic pain 3, and 12 months after cesarean delivery in a cohort of women in University hospital La Paz. We also aim to study the possible contribution of anesthetic and surgical risk factors for the development of Chronic post-surgical pain after cesarean (PCSCP)

DETAILED DESCRIPTION:
* This prospective observational cohort study was conducted at University hospital La Paz. Women hospitalized for cesarean section from March 2017 to September 2018 were recruited on the hospital on the day of surgery, when research interviewers were available. Patients who agreed to participate were interviewed in person preoperatively,at discharge from Reanimation and 24 h postoperatively. Telephone follow-up interviews were conducted one week and 3,and 12 months following surgery. Intraoperative information was collected from the patient record or directly filled by a research person. Questionnaires applied in the present study are reflected in file 1.
* Study participants had to be aged between 18 and 50 years and American Society of Anesthesiologists scale (ASA) had to be I, II or III The exclusion criteria were history of major psychiatric disorder and inability to undertake a personal or telephone interview, ASA> III or dead fetus as result of caesarean section. The study was approved by the local ethics committee (registration number: PI-2564), and written informed consent was obtained from all patients.

Questions about age, race, gestational age, toxic habits, body mass index (BMI) (that was calculated from height and weight) previous vaginal delivery, cesarean delivery, other demographic, medical, surgical, and pre- operative pain variables were included.

-Were also recruited information about urgency level of caesarean using the classification proposed by Lucas et al.use of preoperative oxytocin, anesthesic technique before caesarean section (for example epidural for labor) and surgical and anesthesia variables.

Patients were visited within 24 h after surgery. Pain intensity was assessed as average pain at rest and on movement during the past 24 h using (NRS) and DN2 questionnaire. Also analgesic consumption and relevant side effects or complications were annotated.

Assessment after 3, and 12 months

-Patients were contacted by telephone by one of the authors at 3, and 12 months following cesarean section. This telephone interview usually takes no longer than 15 min. Chronic postsurgical pain (CPSP) was measured using the short form Brief Pain Inventory (BPI) BPI assesses the severity of pain and its impact on functioning. The pain severity items are presented as numeric rating scale (NRS). The patients were asked to rate their pain at rest and during movement in the previous week of the survey. Items of pain interference on function (general activity, mood, walking, work, relations with others, sleep and enjoyment of life ) are also presented as numeric rating scale (NRS) , are valued with 0 = does not interfere and 10 = interferes completely. There were also questions consumption of analgesics and neuropathic pains symptoms using Neuropathic pain (DN2) questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Anesthesiologists scale (ASA) had to be I, II or III

Exclusion Criteria:

* history of major psychiatric disorder and inability to undertake a personal or telephone interview, ASA> III or dead fetus as result of caesarean section

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women hospitalized for cesarean section from March 2017 to September 2018 were recruited on the hospital on the day of surgery. Patients who agreed to participate and meet the inclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 610 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
assess if clinically relevant pain measured by neuropathic pain questionnaire of 2 questions (DN2) > 3/10 one week after cesarean section(CS) was a risk factor for chronic post-surgical pain (CPSP) | three months
  Asses chronic pain 3 months after cesarean delivery in a cohort of women in University Hospital La Paz.A telephone interview with DN2 questionnaire was performed to all patients one week after surgery to assess the presence of neuropathic pain. CPSP diagnosis was retained in patients with the persistence of any symptom of pain or discomfort in the surgical site in the previous week, with an NRS score superior to 3/10 at rest and/or during movement 3 months after surgery.

SECONDARY OUTCOMES:
assess whether a pain intensity superior to 5/10 on the NRS one week after Cesarean Section was related to a higher incidence of CPSP at three months. | Three months
  Asses chronic pain 3 months after cesarean delivery in a cohort of women in University Hospital La Paz. A telephone interview with Numeric Rating Scale (NRS) questionnaire was performed to all patients one week after surgery to assess the presence of moderate pain. (No pain: NRS=0; Mild pain: NRS=1-3; Moderate pain: NRS= 4-6; Severe pain=7-10) CPSP diagnosis was retained in patients with the persistence of any symptom of pain or discomfort in the surgical site in the previous week, with an NRS score superior to 3/10 at rest and/or during movement 3 months after surgery.

OTHER OUTCOMES:
Asses if age of patients, measured as years, is a risk factor for chronic post surgical pain | One week and three months.
  Pain intensity was assessed as average pain at rest and on movement during the past 24 h using NRS and DN2 questionnaire 24 hours, one week and three months after surgery.
Asses if gestational age of patients, measured as week of gestation, is a risk factor for chronic post surgical pain | One week and three months.
  Pain intensity was assessed as average pain at rest and on movement during the past 24 h using NRS and DN2 questionnaire 24 hours, one week and three months after surgery.
Asses if toxic habits of patients, measured as yes/no question: tobacco yes/no and drugs yes/no , is a risk factor for chronic post surgical pain | One week and three months.
  Pain intensity was assessed as average pain at rest and on movement during the past 24 h using NRS and DN2 questionnaire 24 hours, one week and three months after surgery.
Asses if body mass index of patients, measured as kg/ m2, is a risk factor for chronic post surgical pain | One week and three months.
  Pain intensity was assessed as average pain at rest and on movement during the past 24 h using NRS and DN2 questionnaire 24 hours, one week and three months after surgery.
Asses if previous vaginal delivery, measured as yes/no question: previous vaginal delivery yes/no, is a risk factor for chronic post surgical pain. | One week and three months.
  Pain intensity was assessed as average pain at rest and on movement during the past 24 h using NRS and DN2 questionnaire 24 hours, one week and three months after surgery.
Asses if previous cesarean delivery, measured as yes/no question: previous cesarean delivery yes/no, is a risk factor for chronic post surgical pain. | One week and three months.
  Pain intensity was assessed as average pain at rest and on movement during the past 24 h using NRS and DN2 questionnaire 24 hours, one week and three months after surgery.
Asses if previous chronic pelvic pain disorder, measured as a yes/no question: chronic pelvic pain disorder yes/no, is a risk factor for chronic post surgical pain | One week and three months.
  Pain intensity was assessed as average pain at rest and on movement during the past 24 h using NRS and DN2 questionnaire 24 hours, one week and three months after surgery.
Asses if urgency level os cesarean, using classification proposed by lucas et al. is a risk factor for chronic post surgical pain | One week and three months.
  Classification relating the degree of urgency to the presence or absence of maternal or fetal compromise:
  1. Immediate threat to life of woman or fetus
  2. No inmediata threat to life of woman or fetus
  3. Requires early delivery
  4. At a time to suit the woman and maternity services.
  Pain intensity was assessed as average pain at rest and on movement during the past 24 h using NRS and DN2 questionnaire 24 hours, one week and three months after surgery.
Asses if anesthetics technique before cesarean section (epidural for labour) information recruited as yes/no epidural for labour, is a risk factor for chronic post surgical pain | One week and three months.
  Pain intensity was assessed as average pain at rest and on movement during the past 24 h using NRS and DN2 questionnaire 24 hours, one week and three months after surgery.
Asses if preoperative use of oxytocin during labour, information recruited as yes/no use of oxytocin during labour, is a risk factor for chronic post surgical pain. | One week and three months.
  Pain intensity was assessed as average pain at rest and on movement during the past 24 h using NRS and DN2 questionnaire 24 hours, one week and three months after surgery.
Asses if kind of surgical incision: pfannenstiel or vertical is a risk factor for chronic post surgical pain. | One week and three months.
  Pain intensity was assessed as average pain at rest and on movement during the past 24 h using NRS and DN2 questionnaire 24 hours, one week and three months after surgery.
Asses if closure of peritoneum: information recruited as yes/no question: closure of peritoneum yes/no, is a risk factor for chronic post surgical pain. is a risk factor for chronic post surgical pain. | One week and three months.
  Pain intensity was assessed as average pain at rest and on movement during the past 24 h using NRS and DN2 questionnaire 24 hours, one week and three months after surgery.
Asses if closure uterine exteriorization: information recruited as yes/no question: uterine exteriorization yes/no, is a risk factor for chronic post surgical pain. is a risk factor for chronic post surgical pain. | One week and three months.
  Pain intensity was assessed as average pain at rest and on movement during the past 24 h using NRS and DN2 questionnaire 24 hours, one week and three months after surgery.
Asses if duration of surgery (minutes) is a risk factor for chronic post surgical pain. is a risk factor for chronic post surgical pain. | One week and three months.
  Pain intensity was assessed as average pain at rest and on movement during the past 24 h using NRS and DN2 questionnaire 24 hours, one week and three months after surgery.
Asses if anesthesia technique for cesarean section (general, epidural, combined or intradural) is a risk factor for chronic post surgical pain. | One week and three months.
  Pain intensity was assessed as average pain at rest and on movement during the past 24 h using NRS and DN2 questionnaire 24 hours, one week and three months after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Cristina R ROCA, FEA, Principal Investigator — Hospital Universitario La Paz
Locations (1):
- Hospital Universitario La Paz, Madrid, Spain